CLINICAL TRIAL: NCT02841709
Title: Multi-center, Double-blind, Randomized, Placebo-controlled, 5-period, 5-treatment Crossover, Polysomnography Dose-response Study to Assess the Efficacy and Safety of ACT-541468 in Elderly Subjects With Insomnia Disorder
Brief Title: Efficacy and Safety of ACT-541468 in Elderly Subjects With Insomnia Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-078A202
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Insomnia Disorder
Keywords: insomnia; elderly; Polysomnography
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — daridorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Sequence 1 (Experimental): Each subject participates in 5 treatment periods. On the evening of the first 2 days of each period they receive one dose (D) of ACT-541468 or placebo orally in the following order: D4, D2, D3, D1 and P, with D4 = the highest dose (50 mg) and D1 the lowest dose (5 mg). Each treatment period is separated from the next one by a 5- to 12-day washout.
  Interventions: Drug: ACT-541468; Drug: Placebo
- Sequence 2 (Experimental): Each subject participates in 5 treatment periods. On the evening of the first 2 days of each period they receive one dose (D) of ACT-541468 or placebo orally in the following order: D2, P, D4, D3 and D1, with D4 = the highest dose (50 mg) and D1 the lowest dose (5 mg). Each treatment period is separated from the next one by a 5- to 12-day washout.
  Interventions: Drug: ACT-541468; Drug: Placebo
- Sequence 3 (Experimental): Each subject participates in 5 treatment periods. On the evening of the first 2 days of each period they receive one dose (D) of ACT-541468 or placebo orally in the following order: D3, D1, D2, P and D4, with D4 = the highest dose (50 mg) and D1 the lowest dose (5 mg). Each treatment period is separated from the next one by a 5- to 12-day washout.
  Interventions: Drug: ACT-541468; Drug: Placebo
- Sequence 4 (Experimental): Each subject participates in 5 treatment periods. On the evening of the first 2 days of each period they receive one dose (D) of ACT-541468 or placebo orally in the following order: P, D4, D1, D2, D3, with D4 = the highest dose (50 mg) and D1 the lowest dose (5 mg). Each treatment period is separated from the next one by a 5- to 12-day washout.
  Interventions: Drug: ACT-541468; Drug: Placebo
- Sequence 5 (Experimental): Each subject participates in 5 treatment periods. On the evening of the first 2 days of each period they receive one dose (D) of ACT-541468 or placebo orally in the following order: D1, D3, P, D4 and D2 with D4 = the highest dose (50 mg) and D1 the lowest dose (5 mg). Each treatment period is separated from the next one by a 5- to 12-day washout.
  Interventions: Drug: ACT-541468; Drug: Placebo

INTERVENTIONS:
Drug: ACT-541468 — Capsules for oral administration containing ACT-541468 at a strength of 5 mg, 10 mg or 25 mg
Drug: Placebo — Capsules for oral administration matching the ACT-541468 capsules

SUMMARY:
This study evaluates the dose response of ACT-541468 on the change of wake after sleep onset (WASO) assessed by polysomnography (PSG) on the first 2 days of each treatment period.

DETAILED DESCRIPTION:
The study consists of 3 phases: a screening phase, a double-blind treatment phase consisting of 5 periods, and a safety follow-up phase. Safety is monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Male or female aged ≥ 65 years.
* Body mass index (BMI): 18.5 ≤ BMI (kg/m2 ) < 32.0
* Insomnia disorder according to DSM-5 criteria.
* Self-reported history of insufficient sleep quantity.
* Insufficient sleep quantity as collected subjectively in the sleep diary and validated objectively by polysomnography.
* Insomnia Severity Index score ≥ 15.

Exclusion Criteria:

* Any current history of sleep disorder other than insomnia, or any lifetime history of related breathing disorder, periodic limb movement disorder, restless legs syndrome, circadian rhythm disorder, rapid eye movement (REM) behavior disorder, or narcolepsy.
* Self-reported usual daytime napping ≥ 1 hour per day, and ≥ 3 days per week.
* Caffeine consumption ≥ 600 mg per day.
* Shift work within 2 weeks prior to the screening visit, or planned shift work during study.
* Travel ≥ 3 time zones within 1 week prior to the screening visit, or planned travel ≥ 3 time zones during study.
* Hematology or biochemistry test results deviating from the normal range to a clinically relevant extent as per judgment of the Investigator.
* AST and/or ALT > 2 × ULN and/or bilirubin > 1.5 × ULN (except known history of Gilbert's syndrome);
* Severe renal impairment (known or defined as estimated creatinine clearance < 30 mL/min);
* History or clinical evidence of any disease or medical condition or treatment, which may put the subject at risk of participation in the study or may interfere with the study assessments.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (9):
- United States (5):
  - Investigator Site, Brandon, Florida
  - Investigator Site, Chicago, Illinois
  - Investigator Site, Las Vegas, Nevada
  - Investigator Site, New York, New York
  - Investigator Site, Cincinnati, Ohio
- Germany (4):
  - Investigator Site, Berlin
  - Investigator Site, Hamburg
  - Investigator Site, Hanover
  - Investigator Site, Schwerin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zammit G, Dauvilliers Y, Pain S, Sebok Kinter D, Mansour Y, Kunz D. Daridorexant, a new dual orexin receptor antagonist, in elderly subjects with insomnia disorder. Neurology. 2020 May 26;94(21):e2222-e2232. doi: 10.1212/WNL.0000000000009475. Epub 2020 Apr 27. PMID 32341187

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 10 centers in 2 countries (USA and Germany)
Pre-assignment Details: Screening phase: From informed consent to randomization, lasting a max. of 28 days and comprising a screening period (screening visit + at least 7 days at home) and a run-in period (2 consecutive PSG nights on SB placebo, + 5-12 days at home with no treatment). Note: More subjects were randomized (n = 58) than originally planned (n = 50).
Groups:
- Sequence 1 (D4, D2, D3, D1 and P): Each subject participated in 5 treatment periods. On the evening of the first 2 days of each period they received one dose (D) of ACT-541468 or placebo orally in the following order: D4, D2, D3, D1 and P, with D4 = the highest dose (50 mg) and D1 the lowest dose (5 mg). Each treatment period was separated from the next one by a 5- to 12-day washout.
- Sequence 2 (D2, P, D4, D3 and D1): Each subject participated in 5 treatment periods. On the evening of the first 2 days of each period they received one dose (D) of ACT-541468 or placebo orally in the following order: D2, P, D4, D3 and D1, with D4 = the highest dose (50 mg) and D1 the lowest dose (5 mg). Each treatment period was separated from the next one by a 5- to 12-day washout.
- Sequence 3 (D3, D1, D2, P and D4): Each subject participated in 5 treatment periods. On the evening of the first 2 days of each period they received one dose (D) of ACT-541468 or placebo orally in the following order: D3, D1, D2, P and D4, with D4 = the highest dose (50 mg) and D1 the lowest dose (5 mg). Each treatment period was separated from the next one by a 5- to 12-day washout.
- Sequence 4 (P, D4, D1, D2 and D3): Each subject participated in 5 treatment periods. On the evening of the first 2 days of each period they received one dose (D) of ACT-541468 or placebo orally in the following order: P, D4, D1, D2, and D3, with D4 = the highest dose (50 mg) and D1 the lowest dose (5 mg). Each treatment period was separated from the next one by a 5- to 12-day washout.
- Sequence 5 (D1, D3, P, D4 and D2): Each subject participated in 5 treatment periods. On the evening of the first 2 days of each period they received one dose (D) of ACT-541468 or placebo orally in the following order: D1, D3, P, D4 and D2 with D4 = the highest dose (50 mg) and D1 the lowest dose (5 mg). Each treatment period was separated from the next one by a 5- to 12-day washout.
Period: 1st Intervention
Arm/Group | Sequence 1 (D4, D2, D3, D1 and P) | Sequence 2 (D2, P, D4, D3 and D1) | Sequence 3 (D3, D1, D2, P and D4) | Sequence 4 (P, D4, D1, D2 and D3) | Sequence 5 (D1, D3, P, D4 and D2)
Started | 12 | 11 | 12 | 12 | 11
Completed | 12 | 11 | 12 | 12 | 11
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Sequence 1 (D4, D2, D3, D1 and P) | Sequence 2 (D2, P, D4, D3 and D1) | Sequence 3 (D3, D1, D2, P and D4) | Sequence 4 (P, D4, D1, D2 and D3) | Sequence 5 (D1, D3, P, D4 and D2)
Started | 12 | 11 | 12 | 12 | 11
Completed | 12 | 11 | 12 | 12 | 11
Not Completed | 0 | 0 | 0 | 0 | 0
Period: 2nd Intervention
Arm/Group | Sequence 1 (D4, D2, D3, D1 and P) | Sequence 2 (D2, P, D4, D3 and D1) | Sequence 3 (D3, D1, D2, P and D4) | Sequence 4 (P, D4, D1, D2 and D3) | Sequence 5 (D1, D3, P, D4 and D2)
Started | 12 | 11 | 12 | 12 | 11
Completed | 12 | 11 | 12 | 12 | 11
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Sequence 1 (D4, D2, D3, D1 and P) | Sequence 2 (D2, P, D4, D3 and D1) | Sequence 3 (D3, D1, D2, P and D4) | Sequence 4 (P, D4, D1, D2 and D3) | Sequence 5 (D1, D3, P, D4 and D2)
Started | 12 | 11 | 12 | 12 | 11
Completed | 12 | 11 | 12 | 12 | 11
Not Completed | 0 | 0 | 0 | 0 | 0
Period: 3rd Intervention
Arm/Group | Sequence 1 (D4, D2, D3, D1 and P) | Sequence 2 (D2, P, D4, D3 and D1) | Sequence 3 (D3, D1, D2, P and D4) | Sequence 4 (P, D4, D1, D2 and D3) | Sequence 5 (D1, D3, P, D4 and D2)
Started | 12 | 11 | 12 | 12 | 11
Completed | 12 | 11 | 12 | 12 | 11
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3
Arm/Group | Sequence 1 (D4, D2, D3, D1 and P) | Sequence 2 (D2, P, D4, D3 and D1) | Sequence 3 (D3, D1, D2, P and D4) | Sequence 4 (P, D4, D1, D2 and D3) | Sequence 5 (D1, D3, P, D4 and D2)
Started | 12 | 11 | 12 | 12 | 11
Completed | 12 | 11 | 12 | 12 | 11
Not Completed | 0 | 0 | 0 | 0 | 0
Period: 4th Intervention
Arm/Group | Sequence 1 (D4, D2, D3, D1 and P) | Sequence 2 (D2, P, D4, D3 and D1) | Sequence 3 (D3, D1, D2, P and D4) | Sequence 4 (P, D4, D1, D2 and D3) | Sequence 5 (D1, D3, P, D4 and D2)
Started | 12 | 11 | 12 | 12 | 11
Completed | 12 | 11 | 12 | 12 | 11
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Washout Period 4
Arm/Group | Sequence 1 (D4, D2, D3, D1 and P) | Sequence 2 (D2, P, D4, D3 and D1) | Sequence 3 (D3, D1, D2, P and D4) | Sequence 4 (P, D4, D1, D2 and D3) | Sequence 5 (D1, D3, P, D4 and D2)
Started | 12 | 11 | 12 | 12 | 11
Completed | 12 | 11 | 12 | 12 | 11
Not Completed | 0 | 0 | 0 | 0 | 0
Period: 5th Intervention
Arm/Group | Sequence 1 (D4, D2, D3, D1 and P) | Sequence 2 (D2, P, D4, D3 and D1) | Sequence 3 (D3, D1, D2, P and D4) | Sequence 4 (P, D4, D1, D2 and D3) | Sequence 5 (D1, D3, P, D4 and D2)
Started | 12 | 11 | 12 | 12 | 11
Completed | 10 (Note: In total, 2 subjects did not complete Sequence 1.) | 11 | 12 | 12 | 9 (Note: In total, 2 subjects did not complete Sequence 5.)
Not Completed | 2 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Each subject participated in 5 treatment periods. On the evening of the first 2 days of each period they received one dose (D) of ACT-541468 or placebo orally in the following order: D4, D2, D3, D1 and P, with D4 = the highest dose (50 mg) and D1 the lowest dose (5 mg). Each treatment period was separated from the next one by a 5- to 12- day washout.
  ACT-541468: Capsules for oral administration containing ACT-541468 at a strength of 5 mg, 10 mg or 25 mg
  Placebo: Capsules for oral administration matching the ACT-541468 capsules
Arm/Group | All Study Participants
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 57
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 69 [65 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 54
  More than one race | 0
  Unknown or Not Reported | 0
Insomnia Severity Index [Mean (Full Range); unit: units on a scale] — Range 0 - 28.
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
  units on a scale | 20 [15 to 28]

OUTCOME MEASURES:

1. Primary Outcome: Change in Wake After Sleep Onset (WASO) From Baseline to Days 1 and 2
Description: WASO is the time in minutes spent awake after onset of persistent sleep until lights on as determined by polysomnography (PSG)
Time Frame: Baseline to Day 1 and Day 2 of each treatment period
Measure: Least Squares Mean (Standard Error); unit: minutes
Groups:
- ACT-541468 5 mg; ACT-541468 10 mg; ACT-541468 25 mg; ACT-541468 50 mg; Placebo: Each subject participated in 5 treatment periods. On the evening of the first 2 days of each period they received one dose (D) of ACT-541468 or placebo orally in the following order: D4, D2, D3, D1 and P, with D4 = the highest dose (50 mg) and D1 the lowest dose (5 mg). Each treatment period was separated from the next one by a 5- to 12- day washout.
  ACT-541468: Capsules for oral administration containing ACT-541468 at a strength of 5 mg, 10 mg or 25 mg
  Placebo: Capsules for oral administration matching the ACT-541468 capsules
Arm/Group | ACT-541468 5 mg | ACT-541468 10 mg | ACT-541468 25 mg | ACT-541468 50 mg | Placebo
Number analyzed (Participants) | 56 | 54 | 55 | 56 | 54
minutes | -18.9 (4.44) | -32.0 (4.50) | -45.1 (4.47) | -61.4 (4.44) | -13.6 (4.50)
Statistical Analysis 1: Comparison: ACT-541468 5 mg vs ACT-541468 10 mg vs ACT-541468 25 mg vs ACT-541468 50 mg vs Placebo; Multiple Comparison Procedure-Modeling (MCP-Mod) was used to assess a dose response across placebo and all ACT-541468 doses. The null hypothesis of "no dose response" was rejected if at least one of the six Multiple Contrasts Tests (MCTs) had a multiplicity adjusted p-value <0.05. The analysis was performed using the R-package "DoseFinding" (Bornkamp B, Pinheiro J, Bretz F. Planning and analyzing dose finding experiments. 2016. Available from: cranrprojects.org/web/packages/DoseFinding.); Test type: Other; p < 0.001, Multiple Comparison Procedure-Model
Statistical Analysis 2: Comparison: ACT-541468 5 mg vs Placebo; Test type: Other; p = 0.258, Linear mixed effects model; LS mean difference = -5.4, 95% CI 2-sided [-14.7 to 4.0], Standard Error of Mean 4.73 — Parameter Dispersion Type: Standard Error of the LS Mean
Statistical Analysis 3: Comparison: ACT-541468 10 mg vs Placebo; Test type: Other; p < 0.001, Linear mixed effects model; LS mean difference = -18.4, 95% CI 2-sided [-27.8 to -9.0], Standard Error of Mean 4.76 — Parameter Dispersion Type: Standard Error of the LS Mean
Statistical Analysis 4: Comparison: ACT-541468 25 mg vs Placebo; Test type: Other; p < 0.001, Linear mixed effects model; LS mean difference = -31.5, 95% CI 2-sided [-40.9 to -22.2], Standard Error of Mean 4.74
Statistical Analysis 5: Comparison: ACT-541468 50 mg vs Placebo; Test type: Other; p < 0.001, Linear mixed effects model; LS mean difference = -47.8, 95% CI 2-sided [-57.2 to -38.5], Standard Error of Mean 4.74

2. Secondary Outcome: Change in Mean Latency to Persistent Sleep (LPS) From Baseline to Days 1 and 2
Description: LPS is the duration of time in minutes from lights off to persistent sleep onset as determined by PSG
Time Frame: Baseline to Day 1 and Day 2 of each treatment period
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | ACT-541468 5 mg | ACT-541468 10 mg | ACT-541468 25 mg | ACT-541468 50 mg | Placebo
Number analyzed (Participants) | 56 | 54 | 55 | 56 | 54
Minutes | -37.92 (48.76) | -44.61 (41.28) | -44.81 (41.56) | -44.88 (44.22) | -33.88 (41.74)

ADVERSE EVENTS:
Time Frame: Start of screening until the end of the safety follow-up period.
Groups:
- Single-blind Placebo (Run-in Period): Single-blind placebo was administered during the run-in period.
  Placebo: Capsules for oral administration matching the ACT-541468 capsules
- Placebo; ACT-541468 5 mg; ACT-541468 10 mg; ACT-541468 25 mg; ACT-541468 50 mg: Each subject participated in 5 treatment periods. On the evening of the first 2 days of each period they received one dose (D) of ACT-541468 or placebo orally in the following order: D1, D3, P, D4 and D2 with D4 = the highest dose (50 mg) and D1 the lowest dose (5 mg). Each treatment period was separated from the next one by a 5- to 12- day washout.
  ACT-541468: Capsules for oral administration containing ACT-541468 at a strength of 5 mg, 10 mg or 25 mg
  Placebo: Capsules for oral administration matching the ACT-541468 capsules
Arm/Group | Single-blind Placebo (Run-in Period) | Placebo | ACT-541468 5 mg | ACT-541468 10 mg | ACT-541468 25 mg | ACT-541468 50 mg
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/54 | 0/56 | 0/54 | 0/55 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/54 | 0/56 | 0/54 | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 7/58 | 11/54 | 14/56 | 12/54 | 10/55 | 16/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-blind Placebo (Run-in Period) (N=58) | Placebo (N=54) | ACT-541468 5 mg (N=56) | ACT-541468 10 mg (N=54) | ACT-541468 25 mg (N=55) | ACT-541468 50 mg (N=56)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Hyporeflexia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Delusional disorder, unspecified type (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT02841709/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT02841709/SAP_001.pdf